CLINICAL TRIAL: NCT01662154
Title: Percutaneous Nerve Stimulation as a Means to Assess Nerve Block Effectiveness
Brief Title: Neurometer vs Nerve Stimulator: Block Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI no longer at institution
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00031858
Record Dates: First submitted 2012-07-11; First posted 2012-08-10 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Nerve Block Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nerve stimulator (Experimental): Patients in this group will have their nerve blocks assessed with a common nerve stimulator (Stimuplex HNS 12, B.Braun, Germany).
  Interventions: Device: Nerve stimulator assessment
- Neurometer (Active Comparator): Patients in this group will have their nerve block assessed using the Neurometer.
  Interventions: Device: Neurometer assessment

INTERVENTIONS:
Device: Neurometer assessment — Activity of nerve(s) to be blocked will be assessed with the Neurometer before and after administration of local anesthetic.
  Arms: Neurometer
Device: Nerve stimulator assessment — Activity of nerve(s) to be blocked will be assessed with the Stimuplex HNS 12 nerve stimulator before and after administration of local anesthetic.
  Arms: Nerve stimulator

SUMMARY:
Anesthetizing nerves in the extremities is an effective way to freeze an area in preparation for surgery. The doctor injects local anesthetic in an appropriate area, interrupting signals from nerves in that area that control movement and sensation. Depending on how much anesthetic is injected, the doctor can impair both movement and sensation or sensation alone. Currently, there are a few methods used to determine how much sensation a patient has in an area, such as testing the patient's response to a pinprick or cold sensation on the skin. Unfortunately, these methods are subjective and don't always give an accurate measurement of how extensive the block is. For this reason, a more accurate and objective method of assessing nerve blocks is needed. We wish to perform a study to test two nerve stimulation devices to compare their ability to give adequate measurements of nerve activity before and after local anesthesia. If we find that a common nerve stimulator can consistently give accurate readings of nerve activity, anesthesiologists may be able to use this device to determine how well a nerve block is working and adjust the patient's anesthesia accordingly.

DETAILED DESCRIPTION:
Background and rationale Peripheral nerve blocks (PNBs) are highly effective methods of anesthetizing regions of the body for surgery. Throughout its history, the field of regional anesthesiology has lacked an objective, quantitative tool for assessing the effectiveness of a given block. Current methods for assessing blocks are mainly subjective and rely on patient feedback to determine how well a nerve is blocked; these methods include 1) sensory tests, such as ability to detect a pinprick or cold sensation, 2) motor tests, for example, ability to flex or extend the body part that has been blocked, and 3) verbal feedback by the patient. Although these methods usually provide a satisfactory assessment of the block, an objective tool that could decisively and consistently determine how well a nerve is blocked would avoid the ambiguity inherent to the subjective tests and may allow anesthesiologists to more precisely control pain during and after surgery.

Nerve stimulation technology represents one possible method for objectively assessing PNBs by eliciting paresthesia in the region of the body undergoing blockade. Nerve stimulation devices operate by sending an electrical current to a nerve, depolarizing it, and eliciting muscle contraction or paresthesia, depending on the type of nerve stimulated (motor or sensory, respectively). In theory, patients may exhibit a higher current perception threshold in regions of the body that have been anesthetized. Several nerve stimulation devices are commercially available, although they vary in cost, setup, and features. The Neurometer diagnostic stimulator is a percutaneous nerve stimulation device that records sensory nerve conduction thresholds and is commonly used to diagnose neuropathies associated with conditions such as carpal tunnel syndrome, diabetes, and spinal cord lesions. The Neurometer generates constant alternating current sinusoid waveform stimuli at three different calibrated frequencies: 2000 Hz, 250 Hz, and 5 Hz with a range of stimulus output intensities from 0.01 to 9.99 milliAmperes (mA). The current is delivered to the skin surface via a pair of 1 cm diameter gold electrodes separated by 1.7 cm.

Other devices, such as peripheral nerve stimulators, are commonly connected to insulated needles or stimulating catheters to locate nerves to be blocked. When connected to a surface electrode probe, a peripheral nerve stimulator delivers an electric current that elicits motor or sensory activity as the current stimulates the appropriate target nerve. The device generates square pulses with selectable stimulus duration and continuously adjustable stimulation current. The pulse current can be adjusted to appropriate levels, allowing extremely precise adjustments of the stimulation current. The stimulation frequency and stimulus duration can be varied for different applications. The nerve stimulator features the option of selecting a frequency of 1 Hz or 2 Hz for sequential electrical nerve stimulation and stimulus duration of 0.05 milliseconds (ms) to 1 ms.

Although the Neurometer represents the gold standard in percutaneous nerve stimulation, it is expensive, making it impractical for use in everyday clinical applications. We hypothesize that a common peripheral nerve stimulator device can be used as a functional substitute for the Neurometer in generating a sensory stimulus to assess PNB effectiveness. The aim of this study is to compare the Neurometer and a common nerve stimulator to assess anesthesia following PNB. We predict that the nerve stimulator can be used successfully as a substitute for the Neurometer in assessing PNBs in patients receiving regional anesthesia of the extremities.

Study objective To compare the Neurometer and a common peripheral nerve stimulator in measuring current perception threshold in patients receiving PNB.

Hypothesis A nerve stimulator can be used in place of the Neurometer to generate a sensory stimulus to reliably and accurately assess the extent of PNB.

Study procedures This study will recruit patients scheduled for elective surgery at the University of Alberta Hospital (UAH). Since this is an observational study, a sample size of 60 participants will be chosen for convenience. Each week at the UAH, numerous outpatient surgeries are performed on the abdomen and upper and lower extremities, allowing the data to be collected over a span of several months. Potential participants will be recruited by a member of the study team either on the Same-Day Admitting Ward or in the holding area adjacent to the nerve block area and operating theatres. Signed consent will be obtained from each participant; participation will be voluntary and patients have the right to withdraw from the study at any point.

Prior to the nerve block, a member of the study team will record nerve responses in various areas on the patient's extremities (hands, feet) or appropriate sensory area using both the Neurometer and a nerve stimulator (Stimuplex HNS 12, B.Braun, Germany). Common nerve blocks for surgeries of the upper extremities include interscalene, supraclavicular, infraclavicular, while lower extremity surgeries commonly entail spinal or ankle blocks or popliteal blocks of the sciatic nerve. Epidural blocks are commonly used for abdominal surgeries. The Neurometer current perception threshold (CPT) test is administered at standardized cutaneous test sites that are specific for dermatomal and peripheral nerve evaluations. The standardized CPT exam includes preparing each test site with supplied prep paste and testing the subject at each body site with all three frequencies in the following order: 2000 Hz, 250 Hz and 5 Hz. A pair of gold electrodes is coated with a thin layer of conductive gel and then taped to the cutaneous site being tested. Next, an intensity alignment procedure is conducted to approximate the sensory threshold within a 10 mA range. Then, using an automated double-blind (micro-processor controlled) methodology, the subject is presented with 7-10 cycles of randomly selected real and false stimuli, above and below their perception threshold level, until the exact CPT value within that range is determined. This testing methodology is able to determine reproducible CPT measures within a +/-10 mA range. The nerve stimulator test will involve connecting a ground electrode and surface electrode probe (Pajunk, Germany) to the nerve stimulator. The ground electrode will be secured on the body and the current will be delivered by touching the tip of the probe to the same points on the body as tested with the Neurometer. A small amount of conducting gel will be applied to the area to be tested before applying the tip of the probe to the skin. A stimulation frequency of 2 Hz will be used and current will be gradually increased from 0.0 mA until the patient can detect a 'tingling' feeling in the area. The study team will also assess the block using a cold sensation test, in which a cold stimulus (a rubber glove containing ice) is applied to the skin and the patient is asked to give feedback on their perception of the cold stimulus (see below).

After pre-block data has been recorded, patients will receive an ultrasound-guided PNB appropriate to the type of surgery to be performed in standard fashion. After the block has been performed, patients' nerve response in the blocked region will be assessed with the two nerve stimulation devices and the standard cold stimulus test at appropriate intervals (e.g., 10, 20, 30 minutes) until it the patient is ready for surgery. For the electrical stimulus tests, the current required to elicit sensation in the block region at different stimulation frequencies (2 Hz for the nerve stimulator and 2000 Hz, 250 Hz, and 5 Hz for the Neurometer) will be recorded. For the cold stimulus test, a scale measuring sensation will be used (3 = full sensation; 2 = reduced sensation but still cold; 1 = sensation, but not cold; 0 = no sensation). The block will be deemed complete when the current readout on the electrical devices reaches 10 mA and when the cold sensation is 1 or less; at this point, the patient will be transferred to the surgical suite.

Following surgery, patients' nerve response in the blocked region will be assessed with the two devices and the cold stimulus test in the post-anesthesia recovery room. Data will be recorded by hand on data collection sheets and will be transferred to a MS Excel database following the study. Nerve response data obtained with the Neurometer and nerve stimulator will be compared to determine if the nerve stimulator is able to reproduce to a satisfactory extent the nerve stimulation readings of the Neurometer. These results will also be compared to the results of the cold stimulus test to detect any correlation between a patient's nerve response data and when they were able to detect the cold stimulus.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older) patients who have provided informed consent.
* Outpatients scheduled for elective surgery on the upper or lower extremity or abdomen.
* Requirement for nerve block.

Exclusion Criteria:

* Failure to provide informed consent.
* Neuropathic lesions or polyneuropathic conditions.
* Implanted electrical devices (e.g., pacemaker, spinal cord or peripheral nerve stimulator).
* Allergy to local anesthetics.
* Severe coagulopathy.
* Bilateral upper limb surgery.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Accuracy of nerve activity measurement. | During nerve stimulation (approximately 30 seconds for each stimulation test)
  Testing whether a common nerve stimulator device detects nerve activity as accurately and consistently as the Neurometer.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Pither CE, Raj PP, Ford DJ. (1985) The use of peripheral nerve stimulators for regional anesthesia: A review of experimental characteristics, technique, and clinical implications. Reg. Anesth. 10:49-58.
- [Background] Masson EA, Boulton AJ. The Neurometer: validation and comparison with conventional tests for diabetic neuropathy. Diabet Med. 1991;8 Spec No:S63-6. doi: 10.1111/j.1464-5491.1991.tb02159.x. PMID 1825961
- [Background] NEUROMETER® Clinical and Research Update (2010 - 2011). Available at: http://www.neurotron.com/documents_downloads.html
- [Background] Stimuplex® HNS 12 User Manual. B.Braun Melsungen AG. Available at: http://www.bbraun.com/cps/rde/xchg/bbraun-com/hs.xsl/products.html?prid=PRID00001835
- [Background] "Generic IRB Application for Research Involving the Electrodiagnostic sensory Nerve Conduction Threshold (sNCT) Evaluation, August 19, 2004, Diagnostic Transcutaneous Electrical Stimulation in Individuals." Available at: http://www.neurotron.com/documents_downloads.html